CLINICAL TRIAL: NCT05417919
Title: The Effect of Solution-Focused Approach on Attitudes to Violence Against Women in High School Students
Brief Title: Solution-oriented Nursing in Violence Against Women (SONVAW)
Acronym: SONVAW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Principal Investigator, Fatih Sahin, assistant professor, Muş Alparslan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0058
Record Dates: First submitted 2022-06-01; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Violence, Domestic
Keywords: Solution-oriented approach, ,; violence against women,; high school students; psychiatric nurse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Solution-oriented Nursing in Violence Against Women (SONVAW) (Experimental): Initiatives for the Experimental Group Personal Information Form and İSKEBE scale were given to 45 students who were determined in accordance with the research criteria and they were asked to fill in. Data were collected from students who did not come to school that day by telephone or by interviewing them the next day.
  Before the solution-oriented approach program, the students were interviewed and the appropriate time and hours were determined for the program. Then, an online solution-oriented approach program was implemented, which lasted for 6 weeks at the specified hours and days. In the first week of the program, a guide form containing the activities related to the program to be applied was distributed to the students. At the end of the program, the students were asked to fill in the İSKEBE scale as a post-test. Three months after the end of the program, they were asked to fill in the İSKEBE scale again as a follow-up test.
  Interventions: Other: Solution-oriented Nursing in Violence Against Women (SONVAW)
- Control (No Intervention): Initiatives for the Control Group Personal Information Form and İSKEBE scale were given to 45 students who were determined in accordance with the research criteria and they were asked to fill in. Data were collected by phone calls or the next day with students who did not come to school that day. 6 weeks after the pre-test application, the students were asked to fill in the İSKEBE scale as a post-test. Three months after the post-test application, they were asked to fill out the İSKEBE scale again as a follow-up test. At the end of the follow-up test, 45 minutes of violence against women training was given to the control group students.

INTERVENTIONS:
Other: Solution-oriented Nursing in Violence Against Women (SONVAW) — The Personal Information Form was filled in by the students themselves before the program. İSKEBE was filled before, after the program and at the follow-up 3 months later. 3 days were determined for the program for the students in the experimental group, and the program was applied for 60 minutes a day for 6 weeks, allowing the students to participate in the program on a suitable day
  Arms: Solution-oriented Nursing in Violence Against Women (SONVAW)

SUMMARY:
This research was designed as a randomized controlled experimental study with pretest posttest and repeated measurement in order to examine the Effect of Solution-Focused Approach on Attitudes to Violence Against Women in High School Students. The research sample consisted of 90 students (45 control, 45 experiment) who met the inclusion criteria of the research out of 1037 students studying at 5 high schools randomly selected from the central high schools affiliated to the Muş Provincial Directorate of National Education. Personal Information Form and Violence Against Women Attitude Scale (İSKEBE) were used to collect data. The Personal Information Form was filled in by the students themselves before the program. İSKEBE was filled before, after the program and at the follow-up 3 months later. 3 days were determined for the program for the students in the experimental group, and the program was applied for 60 minutes a day for 6 weeks, allowing the students to participate in the program on a suitable day. No intervention was made to the control group during the program. Before the program, the personal characteristics of the control and experimental group students were similar in terms of İSKEBE and subscale scores.

DETAILED DESCRIPTION:
Initiatives for the Experimental Group Personal Information Form and İSKEBE scale were given to 45 students who were determined in accordance with the research criteria and they were asked to fill in. Data were collected from students who did not come to school that day by telephone or by interviewing them the next day. Before the solution-oriented approach program, the students were interviewed and the appropriate time and hours were determined for the program. Then, an online solution-oriented approach program was implemented, which lasted for 6 weeks at the specified hours and days. In the first week of the program, a guide form containing the activities related to the program to be applied was distributed to the students. At the end of the program, the students were asked to fill in the İSKEBE scale as a post-test. Three months after the end of the program, they were asked to fill in the İSKEBE scale again as a follow-up test.

Initiatives for the Control Group Personal Information Form and İSKEBE scale were given to 45 students who were determined in accordance with the research criteria and they were asked to fill in. Data were collected by phone calls or the next day with students who did not come to school that day. 6 weeks after the pre-test application, the students were asked to fill in the İSKEBE scale as a post-test. Three months after the post-test application, they were asked to fill out the İSKEBE scale again as a follow-up test. At the end of the follow-up test, 45 minutes of violence against women training was given to the control group students. During the conduct of the research, both control and experimental group students routinely attended their schools. In addition, no changes were made in the daily life routines of the students.

ELIGIBILITY:
Inclusion Criteria:

* be between the ages of 14-20
* continue high school education
* Not having cognitive, affective and mental limitations
* Not having any problems with hearing and vision skills
* Volunteering to participate in research

Exclusion Criteria:

* failure to meet inclusion criteria

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 78 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
violence against women | before the program
  Before the start of the program, 45 students in the experimental group and 45 students in the control group were given the İSKEBE scale.

SECONDARY OUTCOMES:
violence against women | During the 6-week program
  A solution-oriented approach program was applied to the students who in the experimental group.
violence against women | End of 6-week solution-oriented program
  Immediately after the end of the solution-oriented program, 45 students in the experimental group and 45 students in the control group were given the ISKEBE scale.
violence against women | 3 months after the end of the solution-oriented approach program
  45 students in the experimental group and 45 students in the control group were given the İSKEBE scale.

CONTACTS AND LOCATIONS:
Locations (1):
- MusAlparlanU, Muş, Merkez, Turkey (Türkiye)